CLINICAL TRIAL: NCT04934345
Title: EFFECT OF VASOPRESSORS ON FLUID CHALLENGE PERSISTENCE: AN OBSERVATIONAL STUDY IN PATIENTS UNDERGOING LAPAROTOMY.
Brief Title: EFFECT OF VASOPRESSORS ON FLUID CHALLENGE PERSISTENCE AN OBSERVATIONAL STUDY IN PATIENTS UNDERGOING LAPAROTOMY.
Acronym: NORA_FC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: NORA_FC
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Fluid Challenge; Pharmakodynamic; Norepinephrine; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FC administration: * All the patients receive crystalloids at 4 ml/kg/hour as maintenance fluid during surgery, according to standard practice.
  * After the first episode of hypotension (MAP < 65 mmHg) the PPV is checked.
  * PPV ≥ 13% - FC (4 ml/kg of crystalloids administered in 10')
  * PPV < 13% - start norepinephrine (starting dose - 0.05 mcg/kg/min). In this group, the FC will be administered during an episode of intraoperative hypotension during NE infusion.
  Interventions: Diagnostic Test: Fluid challenge

INTERVENTIONS:
Diagnostic Test: Fluid challenge — The fluid challenge consists of a bolus of 4 ml/kg of crystalloids, administered over 10 minutes.

SUMMARY:
The hemodynamic effect of the fluid challenge administration (FC) depends on different variables related to the interplay between cardiac function and vascular tone response.

In this context, the effect of adding a vasopressor to keep the arterial pressure between predefined ranges may impact on the persistence of stroke volume (SV) changes after FC administration. In fact, both the effect on arterial elastance and venous return may increase the persistence of SV increase, which is know to drop to baseline pre-FC values within fw minutes after FC administration.

This single-centre observational study, in elective patients scheduled for elective laparotomy, hypothesizes that intraoperative norepinephrine infusion would prolong the effect of FC administration.

DETAILED DESCRIPTION:
The appropriate fluid management in the perioperative period is an important, and still partially unclear, chapter of clinical practice for anaesthesiologists. Increasing evidence suggests that intraoperative fluid therapy should be tailored to individual patient's physiology with the purpose of targeting fluid administration to specific stroke volume (SV) responses, or its surrogates. For this reason, small repeated and fast boluses challenging the cardiovascular system should be preferred to continuous and prolonged infusions.

The fluid challenge (FC) is defined as a small amount of fluid given in a short period of time to assess whether the preload reserve of the patient can increase SV with further administration of fluids. A number of studies performed in the operating room evaluated the hemodynamic effects of FC solely considering the effect before and after the infusion. Recently, Aya demonstrated that at least 4 ml kg-1 should be infused to effectively challenge the preload, additionally showing that the hemodynamic effect of the FC is dissipated within 10 minutes, in both responders and in non-responders.

The approach of Aya et al. considers the FC as a drug evoking a systemic response on flow (i.e. SV) and pressure variables [i.e. systolic arterial pressure (SAP)]. Accordingly, the pharmacodynamic effect is evaluated by considering the magnitude (i.e. the maximal changes from baseline obtained for a specific variable), the global effect [i.e. considering the area under the curve (AUC) obtained by plotting the changes overtime] and the persistence of the hemodynamic response after the end of FC administration. The infusion time of FC administration, which ranges in the literature between 5 and 30 minutes, may influence the magnitude of SV response and, in turn, the amount of patients defined as fluid responders . Since several intraoperative pathways of hemodynamic optimization are based on the response to repeated FCs, a prolonged infusion time may potentially affect fluid responsiveness and, in turn, wrongly drive intraoperative fluid management and eventually affect postoperative outcomes.

Since FC is a test embedding at least three variables (i.e. the amount of fluid; the time needed to complete the administration and the SV change threshold used to define a positive response), the role of a one single component on the final outcome can be addressed only by keeping fixed the others. Our group recently investigated the role of the infusion rate in a multicentre study (under revision at the timing of writing this protocol) and our research is now focused on the assessment of the role of the vascular tone in the persistence of the FC effect overtime. The previous study demonstrated that the rate of infusion impact on FC response, however another crucial issue is related to the persistence of the effect of the FC on the SV. In fact, the SV is determined by the interplay between cardiac function and arterial load. Diastolic filling depends on venous return, which is determined by the "stressed volume" and venous compliance. Systolic cardiac function depends on both cardiac factors and arterial load and is predominantly determined by arterial elastance (Ea) and resistance. For this reason, the effect of a vasopressor (i.e. the norepinephrine, the most widely used) may impact on the persistence of the increase of the SV after FC administration.

This single-centre observational study, in elective patients scheduled for elective laparotomy, hypothesizes that intraoperative norepinephrine infusion would prolong the effect of FC administration.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, scheduled for elective laparotomy (>3h predicted) and requiring a FC.

Exclusion Criteria:

* any recurrent cardiac arrhythmia;
* reduced left (ejection fraction < 30%) or right (systolic peak velocity of tricuspid annular motion < 0.17 m/s) ventricular systolic function.

Once enrolled, the patient can be additionally excluded due to the occurrence of one of the following intraoperative conditions:

1. significant bleeding (more than 500 ml in ½ hour)
2. recurrent extrasystoles
3. persistent low quality of the arterial signal affecting hemodynamic monitoring measurements
4. intraoperative hemodynamic instability requiring the persistent use of vasopressors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective surgical patients scheduled for laparotomy >3h
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Stroke volume persistance | evaluated within 10 minutes after fluid challenge infusion
  Stroke volume estimation with respect to baseline values

SECONDARY OUTCOMES:
Pharmakodynamic assesement of FC with and without NE | evaluated within 10 minutes after fluid challenge infusion
  Area under the curve analysis
dmax | evaluated within 10 minutes after fluid challenge infusion
  the maximal percentage difference of the SV observed from baseline
tmax | evaluated within 10 minutes after fluid challenge infusion
  time when dmax maximal value was observed

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Aya HD, Ster IC, Fletcher N, Grounds RM, Rhodes A, Cecconi M. Pharmacodynamic Analysis of a Fluid Challenge. Crit Care Med. 2016 May;44(5):880-91. doi: 10.1097/CCM.0000000000001517. PMID 26683506
- [Background] Vincent JL. Fluid management in the critically ill. Kidney Int. 2019 Jul;96(1):52-57. doi: 10.1016/j.kint.2018.11.047. Epub 2019 Mar 4. PMID 30926137
- [Background] Monnet X, Teboul JL. Assessment of fluid responsiveness: recent advances. Curr Opin Crit Care. 2018 Jun;24(3):190-195. doi: 10.1097/MCC.0000000000000501. PMID 29634494